CLINICAL TRIAL: NCT04165330
Title: A Phase 1/2a Evaluation of the Safety and Efficacy of Adding AL3818 (Catequentinib) to Nivolumab in Solid Tumors
Brief Title: Evaluation of AL3818 in Combination With Nivolumab in Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarcoma Oncology Research Center, LLC (Other)
Collaborators: Advenchen Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL3818-US-005
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor, Adult; Soft Tissue Sarcoma; Non Small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Sarcoma; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — anlotinib; Nivolumab

STUDY DESIGN:
Intervention Model Description: Clinical Trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AL3818 plus nivolumab (Experimental): Part 1: All participants will be assigned to receive AL3818 capsules orally, once daily at sequential deescalating doses (on treatment Days 1-14 followed by no AL3818 treatment from Days 15-21) in combination with nivolumab injection treatment (on Day 1 and Day 15) for a single 21-day cycle. Participants may continue study treatment at the AL3818 cohort dose at investigator discretion.
  Part 2: All participants will receive AL3818 capsules orally, once daily at the RP2D determined from Part 1 (on treatment Days 1-14 followed by no AL3818 treatment from Days 15-21) in combination with nivolumab injection treatment (every 2 weeks starting on Cycle 1, Day 1) in 21-day cycles, for up to 24 cycles of total AL3818 therapy.
  Interventions: Drug: AL3818; Drug: Nivolumab Injection

INTERVENTIONS:
Drug: AL3818 — AL3818: Part 1 - 12 mg, 10 mg, 8 mg, or 6 mg (by dosing cohort), Part 2 - RP2D (as determined from Part 1).
  Administered orally once daily on Days 1-14 per 21 day Cycle.
  Other Names: Anlotinib hydrochloride
Drug: Nivolumab Injection — Nivolumab 240 mg Administered by injection every 2 weeks (Odd Cycles: Days 1 and 15 and Even Cycles Day 8) per 21 day Cycle.
  Other Names: Opdivo

SUMMARY:
This study evaluates the safety and efficacy of AL3818 (anlotinib) hydrochloride in combination with Opdivo (nivilumab) for the treatment patients with of metastatic, advanced, or recurrent solid tumors. All participants will receive open-label AL3818 with nivolumab. Part 1 consists of a dose finding phase to determine the recommended phase 2 dosage of AL3818 with nivolumab. Part 2 consists of a dose expansion phase, evaluating the safety and efficacy of the combination in patients cohorts including metastatic, advanced, or recurrent soft tissue sarcomas, non-small cell lung cancer, and small cell lung cancer.

DETAILED DESCRIPTION:
This phase 1b/2 study evaluates the safety and efficacy of AL3818 (anlotinib) hydrochloride in combination with Opdivo (nivilumab) for the treatment patients with of metastatic, advanced, or recurrent solid tumors including soft tissue sarcomas (STS), non-small cell lung cancer (NSCLC), and small cell lung cancer (SCLC). All participants will receive open-label AL3818 with nivolumab on a scheduled basis.

Part 1 (phase 1b) consists of a dose finding phase to determine the safety, tolerability (including recommended phase 2 dosage (RP2D), and PK profile of AL3818 given with nivolumab. Participants will receive oral AL3818 once daily on Days 1-14 and nivolumab injection on Day 1 and 15 of one 21-day cycle.

Part 2 (phase 2a) consists of a dose expansion phase, to evaluate the safety and preliminary efficacy of combination treatment using AL3818 at the RP2D determined from Part 1 together with nivolumab injection at standard dosing for patients with metastatic, advanced, or recurrent STS, NSCLC, or SCLC in 21-day cycles. Oral AL3818 will be given on Days 1-14 days and nivolumab will be given every 2 weeks, for up to 24 cycles of total AL3818 therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Part 1: Solid tumors of all histologies, including metastatic, locally advanced, or recurrent after at least one prior line of standard therapy and requiring further treatment; OR malignant tumors for which no standard therapy exists, with or without prior therapy.
* Part 2: Histologically confirmed soft tissue sarcomas (STS), small cell lung cancer (SCLC), and non-small cell lung cancer (NSCLC), after at least one prior line of standard therapy and requiring further treatment. For STS subtypes for which no standard therapy exists, patients without prior therapy may be included.
* Measurable disease by RECIST v1.1
* Disease progression or recurrence (after treatment) within 6 months prior to enrollment
* Last dose of prior anti-cancer therapy should be performed at least 21 days prior to the first administration of study treatment.
* Life expectancy of ≥ 3 months at the time of enrollment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Adequate baseline function within 28 days prior to enrollment:

  1. Bone marrow function: Absolute neutrophil count (ANC) ≥ 1,500/mm3; platelets ≥ 100,000/mm3 , Hemoglobin ≥ 9.0 g/dL.
  2. Renal function: Creatinine clearance (calculated by Cockcroft-Gault) must be ≥ 30 ml/min.
  3. Hepatic function: Bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 3.0 x ULN for subjects with Gilbert Syndrome; AST and ALT ≤ 3.0 × ULN.
  4. Coagulation profile: International normalized ratio (INR) is ≤ 2.0; absolute prothrombin time (aPTT) < 1.5 x ULN.
* Left ventricular ejection fraction (LVEF) of > 50% by ECHO or MUGA within 56 days prior to enrollment.
* Two blood pressure readings with systolic blood pressure < 140 mmHg and diastolic blood pressure < 90 mmHg at screening with 28 days prior to enrollment.
* Provide written informed consent before any study-specific procedures are initiated.

Key Exclusion Criteria:

* Major surgical procedure within 28 days or minor surgical procedure within 7 days prior to start of study treatment.
* History of prior or concurrent second primary malignancy that may interfere with the safety or efficacy assessment of the study treatment.
* Untreated, active central nervous system (CNS) metastases.
* Carcinomatous meningitis.
* Active, known, or suspected autoimmune disease or interstitial lung disease.
* Systemic treatment with corticosteroids or other immunosuppressive medications within 14 days prior to start of study treatment.
* Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to start of study treatment.
* History of untreated deep venous thrombosis (DVT) within the past 6 months.
* Presence of uncontrolled infection.
* History of Class III or IV congestive heart failure according to New York Heart Association (NYHA) classification.
* History of any of the following cardiac conditions within 6 months prior to prior to start of study treatment:

  1. Cardiac angioplasty or stenting, or
  2. Myocardial infarction, or
  3. Unstable angina, or
  4. Cerebrovascular accident.
* Presence of any non-healing wound, fracture, or ulcer, or presence of symptomatic peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy or clinically significant bleeding such as gross hematuria, gastrointestinal bleeding and hemoptysis within 6 months prior to start of study treatment.
* QTcF > 470 msec (per Fridericia's formula) on electrocardiogram within 28 prior to start of study treatment.
* Concurrent human Immunodeficiency virus (HIV) infection with CD4+ count < 350 cells/uL.
* Known history of acquired immunodeficiency syndrome (AIDS) and an opportunistic infection within the past 12 months.
* Serologic evidence of chronic hepatitis B virus (HBV) via positive hepatitis B virus surface antigen (HBVsAg) or hepatitis C virus ribonucleic acid (HCV antibody) with a viral load above the limit of quantification.
* History of hepatitis C virus (HCV) infection without completion of curative antiviral treatment with a viral load above the limit of quantification.
* History of organ transplantation.
* Clinical conditions affecting the intake or absorption of AL3818 (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, malabsorption disease, stomach or small bowel resection).
* Known allergies, hypersensitivity, or intolerance to protein-based therapies or with a history of any significant drug allergy (e.g., anaphylaxis, hepatotoxicity, immune-mediated thrombocytopenia or anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) - Part 1 (Phase 1b) | Cycle 1 (21-days)
  Determine the Recommended Phase 2 Dose (RP2D) via evaluation of dose limiting toxicity (DLT) events.
Objective Response Rates (ORR) - Part 2 (Phase 2a) | 18 months
  Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST, v1.1) criteria after three complete 21-day cycles 9 weeks after starting study treatment (C4D1) and then every 12 weeks thereafter for up to C24 cycles. ORR is measured by the number of complete (CR) and partial responses (PR)

SECONDARY OUTCOMES:
Duration of Response (DOR) - Part 2 (Phase 2a) | 30 months
  Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST, v1.1) criteria after three complete 21-day cycles 9 weeks after starting study treatment (C4D1) and then every 12 weeks thereafter for up to C24 cycles. DOR is measured as the median number of months from date of first documented objective response until first documented sign of disease progression or death due to any causes.
Progression Free Survival (PFS) - Part 2 (Phase 2a) | 30 months
  Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST, v1.1) criteria after three complete 21-day cycles 9 weeks after starting study treatment (C4D1) and then every 12 weeks thereafter for up to C24 cycles. PFS is measured as the median number of months from the date of C1D1 until the first documented sign of disease progression or death due to any causes.
Overall Survival (PFS) - Part 2 (Phase 2a) | 30 months
  Evaluated by survival status beginning Cycle 1 Day 1 until last follow up on study. OS is measured as the median number of months from the date of C1D1 until death from any causes.
Clinical Benefit Rate (CBR) - Part 2 (Phase 2a) | 18 months
  Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST, v1.1) criteria after three complete 21-day cycles 9 weeks after starting study treatment (C4D1) and then every 12 weeks thereafter for up to C24 cycles. CBR is measured by the number of CR, PR, and stable diseases (SD).

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events - Parts 1 and 2 | From date of enrollment until final study visit (90 days after last treatment)
  Adverse events and their relationship to study treatment will be assessed at each visit and at unscheduled visits as clinically indicated, according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Sant P Chawla, MD, Principal Investigator — Sarcoma Oncology Research Center
Locations (1):
- Sarcoma Oncology Research Center, Santa Monica, California, United States